CLINICAL TRIAL: NCT07363304
Title: Impact of Elexacaftor-Tezacaftor-Ivacaftor Treatment on Metabolic, Epigenetic and Fecal Microbiota Profiles in People With Cystic Fibrosis.
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Vito Terlizzi, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: MEM-ETI
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Elexacaftor, Tezacaftor, Ivacaftor — Patients with CF, of any age, about to start Elexacaftor, Tezacaftor, Ivacaftor therapy
  Other Names: Trikafta; Kaftrio

SUMMARY:
Cystic Fibrosis (CF) is a genetic disease that affects multiple organs and systems. In recent years, the marketing of CFTR protein modulator drugs, such as the Elexacaftor-Tezacaftor-Ivacaftor (ETI) combination, has significantly improved patients' quality of life and prognosis. ETI, currently prescribed in Italy for CF patients over six years of age with at least one F508del mutation, has shown improvements in lung function, nutritional status, and a reduction in pulmonary exacerbations. In the coming months, ETI will be prescribable for patients aged $\ge$ 2 years with at least one F508del mutation; furthermore, the EMA recently approved its use in all patients aged $\ge$ 2 years, including those with mutations other than F508del (excluding patients with homozygous Class I mutations).Recent studies also highlight an impact on systemic metabolism, with an increase in blood cholesterol levels, blood pressure, and nutritional status, leading to a marked increase in patients with obesity. This could result in an increased long-term cardiovascular risk, especially in children with CF. Additionally, early data show that ETI also induces changes in the gut microbiota and epigenetic modifications by altering DNA methylation, particularly in genes crucial for the onset of CF-related complications, such as diabetes.The gut microbiota of CF patients differs from that of healthy controls, and ETI appears to improve microbial diversity while reducing intestinal inflammation and antibiotic resistance genes. Although ETI-related adverse events are mostly mild and similar to typical respiratory exacerbation symptoms (cough, headache, pharyngodynia, or transient bronchospasm), concerning side effects such as neuropsychiatric effects, intracranial hypertension, or liver failure have also been reported. Currently, it is not possible to predict which patients are at a higher risk of adverse events, but it is known that some of these are related to the blood levels of ETI's individual components. Therefore, monitoring these levels could be useful for dose optimization and reducing the risk of adverse events.Despite the publication of numerous real-world studies on the efficacy and safety of ETI and the sharing of recent standards of care for CF patients on modulator therapy, prospective studies are desirable, especially in the pediatric population. These are needed to monitor metabolic and epigenetic parameters, as well as changes in the fecal microbiota, correlating them with the blood levels of individual ETI components.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF, of any age, about to start ETI therapy, in accordance with marketing authorization Italian legislative directives, followed at the participating CF centers.
* Obtaining informed consent.

Exclusion Criteria:

* CF patients not in ETI therapy and CF patients already in ETI therapy.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll patients with CF pre and post ETI therapy, followed up at included Italian CF centers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in DNA methylation level before and after the start of therapy | baseline, 3, 6, 9, 12, 24 months post-Elexacaftor, Tezacaftor, Ivacaftor

SECONDARY OUTCOMES:
Difference in serum levels of fatty acids, amino acids, sugars and cytokines. | baseline, 3, 6, 9, 12, 24 months post-Elexacaftor, Tezacaftor, Ivacaftor
Correlation between serum levels of fatty acids, amino acids, sugars and cytokines and plasma levels of individual components of the triple modulator therapy (Elexacaftor, Tezacaftor, Ivacaftor) | baseline, 3, 6, 9, 12, 24 months post-Elexacaftor, Tezacaftor, Ivacaftor

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Centro per la Fibrosi Cistica, Azienda Universitaria Ospedaliera Consorziale Policlinico, Bari, Bari
  - Dipartimento di Pediatria, Centro Fibrosi Cistica, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milano
  - Unità Pediatrica, Dipartimento di Scienze Mediche Traslazionali, Centro di Riferimento Regionale per la Fibrosi Cistica, Università degli Studi di Napoli Federico II, Napoli, Napoli
  - Ospedale pediatrico Bambino Gesù, IRCCS, Dipartimento Pediatrico Universitario Ospedaliero, UOC Pneumologia e Fibrosi Cistica, Roma, Roma
  - Centro per la Fibrosi Cistica, Ospedale Infantile Regina Margherita, Torino, Torino
  - Azienda Ospedaliera Universitaria Meyer Istituto di Ricovero e Cura a Carattere Scientifico, Florence

IPD SHARING:
Plan to Share IPD: No